CLINICAL TRIAL: NCT02356965
Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled, Dose Ranging Study to Assess the Analgesic Efficacy, Tolerability, Safety and Pharmacokinetic/Pharmacodynamic Properties of A Sublingual Wafer Formulation of Ketamine Following Third Molar Extraction
Brief Title: Study Testing Ketamine Sublingual Wafer After Wisdom Tooth Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: iX Biopharma Ltd. (Other)
Collaborators: Jean Brown Research (Other); Lotus Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET005
Record Dates: First submitted 2015-01-29; First posted 2015-02-06 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Pain
Keywords: Third molar extraction; Wisdom tooth extraction
MeSH Terms: conditions — Pain | interventions — Ketamine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ketamine 70 mg Sublingual Wafer (Experimental): Single dose of 70 mg ketamine sublingual wafer
  Interventions: Drug: Ketamine
- Ketamine 100 mg Sublingual Wafer (Experimental): Single dose of 100 mg ketamine sublingual wafer
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Single dose of placebo sublingual wafer
  Interventions: Drug: Placebo (for Ketamine)

INTERVENTIONS:
Drug: Ketamine — Single dose of sublingual investigational medication administered when subjects develop moderate to severe pain after third molar extraction.
  Arms: Ketamine 100 mg Sublingual Wafer; Ketamine 70 mg Sublingual Wafer
Drug: Placebo (for Ketamine) — Sublingual sugar pill developed to mimic ketamine sublingual dose.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of the study is to test two different doses of ketamine sub-lingual (under the tongue) wafer against placebo to see how effective the medication is to treat moderate to severe pain after wisdom tooth extraction.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, parallel group, dose-ranging placebo-controlled evaluation of the analgesic efficacy, safety and pharmacokinetics of ketamine sublingual wafer in adult subjects who experience post-operative pain after undergoing third molar extraction.

The study will enroll approximately 80 subjects at a single site. Subjects will be at least 18 years to 38 years of age. Subjects will receive a single dose of 70 mg or 100 mg sublingual ketamine wafer or placebo.

Efficacy assessment will include pain intensity, use of rescue medication, and Patient Global Assessment (PGA) of pain control. Safety assessments will include monitoring of AEs and SAEs, clinical laboratory tests, vital sign measurements, oral assessments, and ECGs.

A maximum of eight 4ml blood samples will be taken from each participant up to 8 hours after study drug administration for plasma analysis.

ELIGIBILITY:
Healthy male and female subjects, ages 18-38 years old, who are scheduled to undergo two ipsilateral third molar extractions.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Sum of Pain Intensity Difference | 3 hours
  Demonstrate the dose-response relationship for analgesia of two dose levels of ketamine sublingual wafer compared with placebo, using the summed pain intensity difference from baseline over the first 3 hours (SPID3) in subjects with acute moderate to severe pain following third molar extraction.

SECONDARY OUTCOMES:
Sum of Pain Intensity Difference | 6 hours
  Summed Pain Intensity Difference at 6 hours (SPID 6).
Safety and Tolerability evaluated by physical examination, vital signs, pulse oximetry, clinical laboratory tests, ECGs and Incident of Adverse Events (AEs) and Serious Adverse Events (SAEs). | 8 hours
  Safety and tolerability of ketamine sublingual wafer as evaluated by physical examination, vital signs, pulse oximetry, clinical laboratory tests, ECGs and Incident of Adverse Events (AEs) and Serious Adverse Events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Derek D Muse, MD, Principal Investigator — Jean Brown Research
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States